CLINICAL TRIAL: NCT06356441
Title: Artificial Intelligence-supported Reading Versus Standard Double Reading for the Interpretation of Magnetic Resonance Imaging in the Detection of Local Recurrence for Nasopharyngeal Carcinoma: a Randomised Controlled Multicenter Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, professor, Sun Yat-sen University
Other Study IDs: B2024-039-01
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Artificial Intelligence Supported Image Reviewing
Keywords: artificial intelligence; image reviewing; magnetic resonance imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI-supported reading: The AI model predicts the incidence of local recurrence. If the incidence is below 60%, one radiologist will interpret the MR images. If the incidence is above 60%, two radiologists will interpret the MR images. The radiologists will be provided with the predictive incidence and contours in their interpretation if desired. If two radiologists provide contradictory interpretations, a third radiologist will participate in the discussion to reach a consensus.
  Interventions: Diagnostic Test: AI
- Standard double reading: The MR images will be interpreted by two radiologists, and in cases of disagreement, a third radiologist will be consulted to reach a consensus.

INTERVENTIONS:
Diagnostic Test: AI — An artificial intelligence model predicts the risk and contours of local recurrence for MR images and triages them before radiologists interpret them.
  Groups: AI-supported reading

SUMMARY:
The aim of this randomized controlled study is to investigate whether the previously developed artificial intelligence model can triage post-radiotherapy magnetic resonance images of patients with nasopharyngeal carcinoma and assist radiologists in their interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with treatment naive nasopharyngeal carcinoma who had finished radiotherapy for 6 months or more
* The previous magnetic resonance imaging examination had showed complete remission in the primary site
* Images are acquired using a 3T magnetic resonance imaging device, including unenhanced T1-weighted and T2-weighted sequences and contrast-enhanced T1-weighted sequences

Exclusion Criteria:

* Patients are enrolled in this study for a specific magnetic resonance imaging scan and not for subsequent follow-up magnetic resonance imaging scans.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study enrolled patients with treatment naive nasopharyngeal carcinoma who have finished radiotherapy for 6 months or more and have no tumor residue in previous examinations.
Sampling Method: Probability Sample
Enrollment: 10400 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
sensitivity | through study completion, an average of 2 years

SECONDARY OUTCOMES:
specificity | through study completion, an average of 2 years
positive predictive value | through study completion, an average of 2 years
negative predictive value | through study completion, an average of 2 years
total time of interpretation for all the MR images | through study completion, an average of 2 years
the rate of discussion with a third radiologist | through study completion, an average of 2 years
the detection rate of local recurrence in the AI-supported reading group | through study completion, an average of 2 years
the sensitivity in the subgroups of different rT-stage | through study completion, an average of 2 years
the incidence of cases whose recurrent risks and contours cannot be provided by the AI model | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Yun Xie, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] OuYang PY, He Y, Guo JG, Liu JN, Wang ZL, Li A, Li J, Yang SS, Zhang X, Fan W, Wu YS, Liu ZQ, Zhang BY, Zhao YN, Gao MY, Zhang WJ, Xie CM, Xie FY. Artificial intelligence aided precise detection of local recurrence on MRI for nasopharyngeal carcinoma: a multicenter cohort study. EClinicalMedicine. 2023 Aug 30;63:102202. doi: 10.1016/j.eclinm.2023.102202. eCollection 2023 Sep. PMID 37680944